CLINICAL TRIAL: NCT00030082
Title: A Phase I Study of Hepatic Arterial Infusion of Escalating Dose Melphalan With Venous Filtration for Metastatic Unresectable Cancers of the Liver
Brief Title: Hepatic Arterial Infusion With Melphalan in Treating Patients With Unresectable Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068941; NCI-01-C-0215; NCT00021606 (obsolete NCT alias)
Record Dates: First submitted 2002-01-30; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2004-07

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Melphalan

INTERVENTIONS:
Drug: isolated perfusion
Drug: melphalan

SUMMARY:
RATIONALE: Heating melphalan to several degrees above body temperature and infusing it to the affected area directly around the tumor may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of hepatic arterial infusion with melphalan in treating patients who have unresectable liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of hepatic arterial infusion with melphalan in patients with unresectable liver cancer.
* Determine the regional and systemic toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients undergo percutaneous hepatic arterial infusion, using a double balloon catheter in the inferior vena cava to isolate circulation to the liver, with melphalan over 30 minutes on day 1. Treatment may be repeated when all toxic effects are grade 2 or less. Patients undergo staging at 4 weeks after completion of the second treatment. Patients may receive 2 additional treatments.

Cohorts of 3-6 patients receive escalating doses of melphalan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 12 additional patients are treated with melphalan at the recommended dose.

Patients are followed every 3 months for 2 years and then every 4 months for 1 year.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable cancer of the parenchyma of the liver
* Liver metastases allowed
* Limited unresectable extrahepatic disease (including but not limited to the following) is allowed provided the life-threatening component of progressive disease is in liver:

  * Up to 4 pulmonary nodules each less than 1 cm in diameter
  * Retroperitoneal lymph nodes less than 3 cm in diameter
  * Fewer than 10 skin or subcutaneous metastases less than 1 cm in diameter
  * Asymptomatic bone metastases that have been or can be palliated with radiotherapy
  * Solitary metastasis to any site that can be resected
* Prior therapy with intrahepatic perfusion with or without hepatic arterial infusion with floxuridine is allowed provided patient had a radiographic partial response of 3-months duration

PATIENT CHARACTERISTICS:

Age:

* 14 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Absolute neutrophil count at least 1,300/mm^3
* Hematocrit greater than 27%

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* PT within 2 seconds of upper limit of normal
* No biopsy-proven cirrhosis with evidence of portal hypertension by history, endoscopy, or radiologic study

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No prior congestive heart failure with LVEF less than 40%

Pulmonary:

* No chronic obstructive pulmonary disease
* No other chronic pulmonary disease
* FEV_1 at least 30% of predicted
* DLCO at least 40% of predicted

Other:

* Weight greater than 35 kg
* HIV negative
* No active infections
* No severe allergic reaction to iodine contrast not controlled by antihistamines or steroids
* No known prior hypersensitivity reaction to melphalan
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 month since prior biologic therapy for the malignancy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 1 month since prior chemotherapy for the malignancy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 1 month since prior radiotherapy for the malignancy and recovered

Surgery:

* Not specified

Other:

* No concurrent chronic anticoagulants
* No concurrent immunosuppressive drugs

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Alexander, MD, FACS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States